CLINICAL TRIAL: NCT01316341
Title: Pharmacokinetics and Pharmacodynamics of BI 10773 After Single and Multiple Oral Dose of 10 mg and 25 mg BI 10773 in Chinese Male and Female Type 2 Diabetic Patients
Brief Title: Pharmacokinetics, Pharmacodynamics, Safety, and Tolerability of Empagliflozin in Chinese Female and Male Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1245.44
Record Dates: First submitted 2011-03-15; First posted 2011-03-16 (Estimated); Results first posted 2014-06-17 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin

ARMS (3):
- BI10773 low dose Per Os(p.o.) (Experimental): patient to receive a tablet containing low dose BI10773 Per Os(p.o.) plus one placebo
  Interventions: Drug: Placebo; Drug: BI10773
- Placebo (Placebo Comparator): patient to receive two placebos
  Interventions: Drug: Placebo
- BI10773 high dose Per Os(p.o.) (Experimental): patient to receive a tablet containing high dose BI10773 Per Os(p.o.) plus one placebo
  Interventions: Drug: BI10773; Drug: Placebo

INTERVENTIONS:
Drug: BI10773 — patient to receive a tablet containing high dose BI10773 p.o. plus one placebo
  Arms: BI10773 high dose Per Os(p.o.)
Drug: Placebo — patient to receive two placebos
  Arms: Placebo
Drug: Placebo — patient to receive two placebos
  Arms: BI10773 low dose Per Os(p.o.)
Drug: Placebo — patient to receive two placebos
  Arms: BI10773 high dose Per Os(p.o.)
Drug: BI10773 — patient to receive a tablet containing low dose BI10773 p.o. plus one placebo
  Arms: BI10773 low dose Per Os(p.o.)

SUMMARY:
the pharmacokinetics, pharmacodynamics and safety and tolerability of single and multiple oral doses of BI 10773 at low dose once daily (q.d.) and high dose q.d. administered to Chinese female and male patients with type 2 diabetes will be investigated.

ELIGIBILITY:
Inclusion criteria:

1. Chinese male and female patients with proven diagnosis of type 2 diabetes mellitus treated with diet and exercise only or on a maximum of two oral antidiabetic agents except thiazolidinediones with at least one agent taken at 50% of its maximum dose or less, unchanged for at least 12 weeks before randomization
2. Glycosylated haemoglobin A1(HbA1c)<=8.5% and >=7.0% at screening,age>=21 and age<=70 years (male and female patients),BMI>=19 and <=40 kg/m2
3. Signed and dated written informed consent by date of Visit 1 in accordance with GCP and local legislation.

Exclusion criteria:

1. Patient who did not discontinue the antidiabetic treatment with insulin or glitazones, DPP-IV at least before 12 weeks before randomization
2. Uncontrolled hyperglycaemia with a glucose level >240 mg/dl (>13.3 mmol/L) after an overnight fast at screening visit
3. Clinically relevant concomitant diseases other than type 2 diabetes, hyperlipidaemia and medically treated hypertension, such as:

4 Any late stage complication of diabetes (e.g. retinopathy, polyneuropathy, vegetative disorders, diabetic foot) 5 Renal insufficiency (calculated creatinine clearance < 80 ml/min/1.73m²) 6 Cardiac insufficiency NYHA II-IV, myocardial infarction, other known cardiovascular diseases including hypertension > 160/95mmHg (measured at training visit and each of the timepoints of Day -1), stroke and TIA 7 Neurological disorders (such as epilepsy) or psychiatric disorders 8 Acute or relevant chronic infections (e.g. HIV, repeated urogenital infections) 9 Any gastrointestinal, hepatic, respiratory, endocrine or immunological disorder 10. History of relevant allergy/hypersensitivity (including allergy to drug or its excipients) 11. A marked baseline prolongation of QT/QTc interval (e.g., ECG demonstration of a QTc interval >450 ms ) at screening visit

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-03; Primary Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1245.44.86001 Boehringer Ingelheim Investigational Site, Beijing, China

REFERENCES:
- [Derived] Zhao X, Cui Y, Zhao S, Lang B, Broedl UC, Salsali A, Pinnetti S, Macha S. Pharmacokinetic and Pharmacodynamic Properties and Tolerability of Single- and multiple-dose Once-daily Empagliflozin, a Sodium Glucose Cotransporter 2 Inhibitor, in Chinese Patients With Type 2 Diabetes Mellitus. Clin Ther. 2015 Jul 1;37(7):1493-502. doi: 10.1016/j.clinthera.2015.05.001. Epub 2015 Jun 19. PMID 26101175

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Two placebo tablets, one matching the empa 10mg tablet and one matching the empa 25mg tablet, taken orally either as a single dose (single dose period) or for 7 consecutive days (multiple dose period).
- Empa 10 mg: 10 mg Empagliflozin (empa) taken orally either as a single dose (single dose period) or for 7 consecutive days (multiple dose period). Along with this a placebo tablet matching the 25mg empa tablet was taken at each drug administration.
- Empa 25 mg: 25 mg Empagliflozin (empa) taken orally either as a single dose (single dose period) or for 7 consecutive days (multiple dose period). Along with this a placebo tablet matching the 10mg empa tablet was taken at each drug administration.
Period: Overall Study
Arm/Group | Placebo | Empa 10 mg | Empa 25 mg
Started | 6 | 9 | 9
Completed | 6 | 9 | 9
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Empa 10 mg | Empa 25 mg | Total
Number analyzed (Participants) | 6 | 9 | 9 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.5 (9.6) | 54.1 (7.9) | 52.7 (9.9) | 53.4 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 6 | 10
  Male | 4 | 7 | 3 | 14

OUTCOME MEASURES:

1. Primary Outcome: Maximum Measured Concentration (Cmax)
Description: Maximum measured concentration of the analyte in plasma after the first dose on day 1.
Time Frame: 5 minutes (min) before drug administration and 10 min, 20min, 30min, 40min, 1 hour (h), 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 12h, 16h after drug administration
Population: Pharmacokinetic (PK) analysis set included all evaluable patients documented to have taken at least one dose of investigational treatment and who provided at least one observation for at least one PK endpoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Groups:
- Empa 10 mg: 10 mg empagliflozin (empa) taken orally as a single dose, plus a placebo tablet matching the 25mg empa tablet.
- Empa 25 mg: 25 mg empagliflozin (empa) taken orally as a single dose, plus a placebo tablet matching the 10mg empa tablet.
Arm/Group | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 9 | 9
nmol/L | 436 (14.1) | 1090 (29.2)

2. Primary Outcome: Time to Maximum Measured Concentration (Tmax)
Description: Time from dosing to the maximum measured concentration of the analyte in plasma, after the first dose on day 1.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 9 | 9
hours | 1.13 (33.3) | 1.50 (40.8)

3. Primary Outcome: Area Under the Curve 0 to Infinity (AUC0-∞) After Single Dosing
Description: Area under the concentration-time curve of empagliflozin (empa) in plasma over the time interval from 0 extrapolated to infinity, after the first dose on day 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 9 | 9
nmol*h/L | 2560 (12.3) | 7250 (24.4)

4. Primary Outcome: Area Under the Curve 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of empagliflozin (empa) in plasma over the time interval from 0 to the time of the last quantifiable data point, after the first dose on day 1.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 9 | 9
nmol*h/L | 2510 (12.3) | 7070 (24.1)

5. Primary Outcome: Terminal Rate Constant (λz)
Description: Terminal Rate Constant in Plasma (λz), after the first dose on day 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/h
Arm/Group | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 9 | 9
1/h | 0.0749 (30.3) | 0.0664 (22.2)

6. Primary Outcome: Terminal Half-life (t1/2)
Description: Terminal half-life of empagliflozin (empa) in plasma after the first dose on day 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 9 | 9
hours | 9.25 (30.3) | 10.4 (22.2)

7. Primary Outcome: Mean Residence Time (MRTpo)
Description: Mean residence time of empagliflozin (empa) in the body after the first dose on day 1.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 9 | 9
hours | 9.29 (16.4) | 10.2 (13.2)

8. Primary Outcome: Apparent Clearance of Empagliflozin After Extravascular Administration (CL/F)
Description: Apparent clearance of empagliflozin (empa) in plasma after extravascular administration, after the first dose on day 1.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 9 | 9
mL/min | 144 (12.3) | 127 (24.4)

9. Primary Outcome: Apparent Volume of Distribution During the Terminal Phase λz (Vz/F)
Description: Apparent volume of distribution during the terminal phase λz, after the first dose on day 1.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 9 | 9
L | 115 (31.8) | 115 (30.1)

10. Primary Outcome: Amount of Empagliflozin Eliminated in Urine in the Time Interval 0 Hours to 24 Hours (Ae 0-24)
Description: Amount of empagliflozin (empa) eliminated in urine in the time interval 0 hours to 24 hours, after the first dose on day 1.
Time Frame: Sampling intervals were 0-2 hours (h), 2-4h, 4-8h, 8-12h and 12-24h after drug administration
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol
Arm/Group | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 9 | 9
nmol | 4030 (18.9) | 9940 (23.8)

11. Primary Outcome: Fraction of Empagliflozin Excreted Unchanged in Urine in the Time Interval 0 Hours to 24 Hours (fe 0-24).
Description: Fraction of empagliflozin (empa) excreted unchanged in urine in the time interval 0 hours to 24 hours, after the first dose on day 1.
Time Frame: Sampling intervals were 0-2 hours (h), 2-4h, 4-8h, 8-12h and 12-24h after drug administration
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of empa
Arm/Group | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 9 | 9
percentage of empa | 18.2 (18.9) | 17.9 (23.8)

12. Primary Outcome: Renal Clearance After Extravascular Administration (CL R,0-48)
Description: Renal clearance of empagliflozin (empa) in plasma after extravascular administration, after the first dose on day 1.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 9 | 9
mL/min | 28.9 (22.6) | 25.6 (31.8)

13. Primary Outcome: Maximum Measured Concentration Over a Uniform Dosing Interval (Cmax,ss)
Description: Maximum measured concentration of empagliflozin (empa) in plasma at steady state over a uniform dosing interval.
Time Frame: 5 minutes (min) before drug administration and 10min, 20min, 30min, 40min, 1 hour (h), 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 12h, 16h, 24h, 36h 48h, 60h, 72h and 96h after drug administration on day 9
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Groups:
- Empa 10 mg: 10 mg empagliflozin (empa) taken orally once daily for 7 consecutive days, plus a placebo tablet matching the 25mg empa tablet taken at each drug administration.
- Empa 25 mg: 25 mg empagliflozin (empa) taken orally once daily for 7 consecutive days, plus a placebo tablet matching the 10mg empa tablet taken at each drug administration.
Arm/Group | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 9 | 9
nmol/L | 489 (27.4) | 1250 (32.1)

14. Primary Outcome: Time From Last Dosing to Maximum Measured Concentration Over a Uniform Dosing Interval at Steady State (Tmax,ss)
Description: Time from last dosing to maximum measured concentration of empagliflozin (empa) in plasma over a uniform dosing interval at steady state, after multiple dosing.
Time Frame: as for outcome 13
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 9 | 9
hours | 1.17 (43.8) | 1.37 (35.0)

15. Primary Outcome: Area Under the Concentration-time Curve in Plasma at Steady State Over a Uniform Dosing Interval (AUCτ,ss)
Description: Area under the concentration-time curve of empagliflozin (empa) in plasma at steady state over a uniform dosing interval, after multiple dosing
Time Frame: as for outcome 13
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 9 | 9
nmol*h/L | 2650 (15.4) | 7520 (21.4)

16. Primary Outcome: Terminal Rate Constant in Plasma at Steady State (λz,ss)
Description: Terminal rate constant in plasma at steady state, after multiple dosing.
Time Frame: as for outcome 13
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/h
Arm/Group | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 9 | 9
1/h | 0.0559 (52.5) | 0.0588 (24.6)

17. Primary Outcome: Terminal Half-life in Plasma at Steady State (t1/2,ss)
Description: Terminal half-life of empagliflozin (empa) in plasma at steady state, after multiple dosing.
Time Frame: as for outcome 13
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 9 | 9
hours | 12.4 (52.5) | 11.8 (24.6)

18. Primary Outcome: Mean Residence Time at Steady State (MRTpo,ss)
Description: Mean residence time of empagliflozin (empa) in the body at steady state after multiple oral administrations
Time Frame: as for outcome 13
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 9 | 9
hours | 10.5 (18.5) | 10.2 (19.1)

19. Primary Outcome: Apparent Clearance of Empagliflozin After Extravascular Administration (CL/Fss)
Description: Apparent clearance of empagliflozin (empa) in the plasma at steady state following multiple oral dose administration.
Time Frame: as for outcome 13
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 9 | 9
mL/min | 139 (15.4) | 123 (21.4)

20. Primary Outcome: Apparent Volume of Distribution During the Terminal Phase λz (Vz/Fss)
Description: Apparent volume of distribution during the terminal phase λz at steady state following oral administration after multiple dosing
Time Frame: as for outcome 13
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 9 | 9
L | 150 (55.1) | 125 (29.9)

21. Primary Outcome: Amount of Analyte Eliminated in Urine at Steady State in Time Interval 0 Hours to 24 Hours (Ae 0-24,ss)
Description: Amount of empagliflozin (empa) eliminated in urine at steady state in the time interval 0 hours to 24 hours, after multiple dosing.
Time Frame: Sampling intervals were 0-2 hours (h), 2-4h, 4-8h, 8-12h and 12-24h after drug administration
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol
Arm/Group | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 9 | 9
nmol | 4420 (14.6) | 11600 (23.3)

22. Primary Outcome: Fraction of Empagliflozin Excreted Unchanged in Urine at Steady State in the Time Interval 0 Hours to 24 Hours (fe 0-24,ss)
Description: Fraction of empagliflozin (empa) excreted unchanged in urine at steady state in the time interval 0 hours to 24 hours, after multiple dosing.
Time Frame: Sampling intervals were 0-2 hours (h), 2-4h, 4-8h, 8-12h and 12-24h after drug administration
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of empa
Arm/Group | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 9 | 9
percentage of empa | 19.9 (14.6) | 20.9 (23.3)

23. Primary Outcome: Renal Clearance at Steady State (CL R,ss)
Description: Renal clearance of empagliflozin (empa) in plasma after extravascular administration, after multiple dosing.
Time Frame: as for outcome 13
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 9 | 9
mL/min | 27.8 (15.8) | 26.1 (30.0)

24. Primary Outcome: Accumulation Ratio Based on AUC (R A,AUC)
Description: Accumulation ratio of empagliflozin (empa) based on AUC, after multiple dosing
Time Frame: 5 minutes (min) before drug administration and 10min, 20min, 30min, 40min, 1 hour (h), 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 12h, and16h after drug administration on days 1 and 9
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 9 | 9
Ratio | 1.14 (12.0) | 1.17 (11.2)

25. Primary Outcome: Accumulation Ratio Based on Cmax (R A,Cmax)
Description: Accumulation ratio of empagliflozin (empa) based on Cmax, after multiple dosing
Time Frame: 5 minutes (min) before drug administration and 10min, 20min, 30min, 40min, 1 hour (h), 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 12h, and16h after drug administration between days 5 and 9
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 9 | 9
Ratio | 1.12 (32.0) | 1.15 (30.8)

26. Primary Outcome: Predose Plasma Concentration Before Planned Dose x (Cpre,x)
Description: Predose plasma concentration of empagliflozin (empa) before planned dose by day.
  This endpoint in steady state is identical to Cmin,ss.
Time Frame: 5 minutes before drug administration
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Groups:
- Empa 10 mg: A single dose of 10 mg Empagliflozin (empa) taken orally, plus one placebo tablet.
- Empa 25 mg: A single dose of 25 mg empagliflozin (empa) taken orally, plus one placebo tablet.
Arm/Group | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 9 | 9
nmol/L
  Treatment Day 5 | 24.64 (1.24) | 70.54 (1.48)
  Treatment Day 6 | 25.70 (1.23) | 80.27 (1.42)
  Treatment Day 7 | 25.24 (1.24) | 78.96 (1.57)
  Treatment Day 8 | 26.10 (1.22) | 72.74 (1.43)
  Treatment Day 9 | 27.21 (1.23) | 76.02 (1.42)

27. Secondary Outcome: Clinical Relevant Abnormalities for Protocol-Specified Significant Adverse Events, Hypoglycaemic Events, Vital Signs, Blood Chemistry, Rescue Therapy, Body Weight and Waist Circumference
Description: Clinically relevant abnormalities for protocol-specified significant adverse events, hypoglycaemic events, vital signs, blood chemistry, use of rescue therapy, change in body weight and change in waist circumference.
  Results shown are for hypoglycaemic events, as this was the only event that occurred for this endpoint.
Time Frame: Drug administration until end of trial, up to 21 days
Population: Treated set (TS) includes all patients who were documented to have taken at least one dose of investigational treatment.
Measure: Number; unit: participants
Arm/Group | Placebo | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 6 | 9 | 9
participants | 0 | 1 | 0

28. Primary Outcome: Urinary Glucose Excretion (UGE) Change From Baseline
Description: Change from day -1 in urinary glucose excretion in a 24 hour collection period per time point.
Time Frame: Sampling intervals were 0-2 hours (h), 2-4h, 4-8h, 8-12h and 12-24h after drug administration
Population: Pharmacodynamic analysis (PD) set included all patients documented to have taken at least one dose of investigational treatment, who received at least one dose of empagliflozin or placebo and who provided at least one baseline and post-treatment observation for at least one PD endpoint.
Measure: Mean (Standard Deviation); unit: mg
Groups:
- Placebo: Two placebo tablets, one matching the empa 10mg tablet and one matching the empa 25mg tablet, taken orally for 7 consecutive days.
Arm/Group | Placebo | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 6 | 9 | 9
mg
  Day 1 | -988.38 (2791.68) | 87680.85 (22924.91) | 82791.86 (18752.81)
  Day 9 | -4106.10 (6428.12) | 95765.72 (24133.47) | 82633.88 (34757.02)

29. Primary Outcome: Fasting Plasma Glucose (FPG) Change From Baseline
Description: Fasting Plasma Glucose (FPG) change from baseline between day 1 and day 9.
Time Frame: Sampling intervals were 0-2 hours (h), 2-4h, 4-8h, 8-12h and 12-24h after drug administration
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Empa 10 mg | Empa 25 mg
Number analyzed (Participants) | 6 | 9 | 9
mg/dL | -3.67 (7.45) | -25.56 (20.74) | -31.44 (26.92)

ADVERSE EVENTS:
Time Frame: Drug administration until end of trial, up to 21 days
Arm/Group | Placebo | Empa 10 mg | Empa 25 mg
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 3/6 | 4/9 | 2/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=6) | Empa 10 mg (N=9) | Empa 25 mg (N=9)
White blood cell disorder (Blood and lymphatic system disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 2 | 1
Eosinophil count abnormal (Investigations) | 1 | 0 | 0
Neutrophil count abnormal (Investigations) | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.